CLINICAL TRIAL: NCT02658331
Title: Clinical Evaluation of the BioFire FilmArray® BioThreat-E Test for the Diagnosis of Ebola Virus Disease in West Africa
Brief Title: Evaluation of the FilmArray BioThreat-E Test
Status: Completed | Type: Observational
Sponsor: BioMérieux (Industry)
Collaborators: Fondation Mérieux (Other); Donka University Hospital, Conakry (Unknown)
Responsible Party: Sponsor
Other Study IDs: EbolaFire
Record Dates: First submitted 2016-01-06; First posted 2016-01-18 (Estimated); Last update posted 2016-01-18 (Estimated); Status verified 2016-01

CONDITIONS: Ebola Virus Disease
Keywords: Ebola Virus Disease; Rapid Diagnosis; Point of care; Molecular platform
MeSH Terms: conditions — Hemorrhagic Fever, Ebola

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood Urine Saliva
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of our study is to assess the analytical and clinical performance of the FilmArray (FA) BioThreat-E test (BioFire®) for the diagnosis of Ebola virus disease in the field in Guinea versus conventional molecular techniques.

DETAILED DESCRIPTION:
The study will be conducted at the "Laboratoire des Fièvres Hémorragiques Virales" in Donka National Hospital (Conakry, Guinea), which is the Reference Laboratory for Hemorrhagic Fevers in Guinea. The reference based population includes the regions of Conakry and Coyah. No specific invasive intervention is required for this research protocol and the study does not interfere with the management of the patients according to the ongoing practices in Donka Ebola Treatment Center and in Coyah Ebola Treatment Center. Each participant will be verbally informed before signing an informed consent. Clinical data will be collected and recorded via a source document questionnaire - Clinical Report Form - based on the routine clinical data already provided to the laboratory according to the practices. Another questionnaire will be submitted to the biologist and technicians involved in the study to assess the practicability of the FilmArray technology, compared to conventional techniques, in terms of time to results, duration of test manipulation, sense of personnel safety for specimen handling, overall workload after each day, and preference of lab professionals.

As the main objective, analytical performance (sensitivity and specificity) and clinical performance (positive and negative predictive values) of the FA BioThreat-E test in whole blood will be evaluated in comparison with the QuantiTect® Probe RT-PCR (Qiagen) and the RealStar® Filovirus Type RT-PCR Kit 1.0 (Altona) both tests performed on serum.

The status for EVD will be defined for each patient based on the result of routine testing:

* Positive patients: patients enrolled in the study showing positive results with the two routine PCR performed in the lab: QuantiTect Probe RT-PCR® and RealStar® Filovirus Type RT-PCR Kit 1.0.
* Negative patients: patients enrolled in the study showing negative results with the two routine PCR performed in the lab: QuantiTect Probe RT-PCR® and RealStar® Filovirus Type RT-PCR Kit 1.0.
* Equivocal patients: all other results showing a discrepancy between the two routine tests.

As a secondary objective, the possibility of using the FilmArray (FA) BioThreat-E test on non-invasive specimens will also be assessed. Urine and saliva specimens will be analyzed by FA for confirmed positive cases only (based on routine testing), for patients able to provide saliva and/or urine specimens according to their health condition.

This research protocol was approved by the Guinean Ethical Committee.

ELIGIBILITY:
Inclusion Criteria:

* All patients, male and female, older than 18, sent to Conakry or Coyah Ebola Treatment Centers for a suspicion of EVD according to WHO criteria, and considered as eligible for Ebola routine diagnosis.
* Ability to deliver a written informed consent

Exclusion Criteria:

* Age below 18.
* Inability to provide a consent
* Inability to provide the blood specimens required for Ebola virus disease diagnosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients, male and female, older than 18, sent to Conakry or Coyah Ebola Treatment Centers for a suspicion of Ebola Virus Disease according to WHO criteria, and considered as eligible for Ebola routine diagnosis.
Sampling Method: Probability Sample
Enrollment: 156 (Actual)
Dates: Start 2015-03; Primary Completion 2015-07 (Actual); Study Completion 2015-07 (Actual)

PRIMARY OUTCOMES:
Number of positive/negative patients for the detection of Ebola virus RNA with the BioThreat-E test performed on whole blood. | Through study completion, an average of 6 months.
  Number of positive/negative patients for the detection of Ebola virus RNA with the BioThreat-E test in comparision with their Ebola Virus Disease status as defined based on the result of routine testing.

SECONDARY OUTCOMES:
Number of urine specimens positive/negative for the detection of Ebola virus RNA with the BioThreat-E test, in patients positive for Ebola Virus Disease based on routine testing, and able to provide a urine specimen. | Through study completion, an average of 6 months.
Number of saliva specimens positive/negative for the detection of Ebola virus RNA with the BioThreat-E test, in patients positive for Ebola Virus Disease based on routine testing, and able to provide a saliva specimen. | Through study completion, an average of 6 months.

CONTACTS AND LOCATIONS:
Overall Officials: Françoise Gay-Andrieu, MD-PhD, Study Chair — BioMérieux; N'Fally Magassouba, PhD, Principal Investigator — Laboratoire des Fièvres Hémorragiques en Guinée - Université Gamal Nasser, Conakry.; Mark Miller, MD-FRCPC, Study Director — BioMérieux

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Leski TA, Ansumana R, Taitt CR, Lamin JM, Bangura U, Lahai J, Mbayo G, Kanneh MB, Bawo B, Bockarie AS, Scullion M, Phillips CL, Horner CP, Jacobsen KH, Stenger DA. Use of the FilmArray System for Detection of Zaire ebolavirus in a Small Hospital in Bo, Sierra Leone. J Clin Microbiol. 2015 Jul;53(7):2368-70. doi: 10.1128/JCM.00527-15. Epub 2015 May 13. PMID 25972415
- [Background] Southern TR, Racsa LD, Albarino CG, Fey PD, Hinrichs SH, Murphy CN, Herrera VL, Sambol AR, Hill CE, Ryan EL, Kraft CS, Campbell S, Sealy TK, Schuh A, Ritchie JC, Lyon GM 3rd, Mehta AK, Varkey JB, Ribner BS, Brantly KP, Stroher U, Iwen PC, Burd EM. Comparison of FilmArray and Quantitative Real-Time Reverse Transcriptase PCR for Detection of Zaire Ebolavirus from Contrived and Clinical Specimens. J Clin Microbiol. 2015 Sep;53(9):2956-60. doi: 10.1128/JCM.01317-15. Epub 2015 Jul 8. PMID 26157148
- [Background] Weller SA, Bailey D, Matthews S, Lumley S, Sweed A, Ready D, Eltringham G, Richards J, Vipond R, Lukaszewski R, Payne PM, Aarons E, Simpson AJ, Hutley EJ, Brooks T. Evaluation of the Biofire FilmArray BioThreat-E Test (v2.5) for Rapid Identification of Ebola Virus Disease in Heat-Treated Blood Samples Obtained in Sierra Leone and the United Kingdom. J Clin Microbiol. 2016 Jan;54(1):114-9. doi: 10.1128/JCM.02287-15. Epub 2015 Nov 4. PMID 26537445